CLINICAL TRIAL: NCT04814147
Title: Role of NLRP3 Inflammasome Activation of Adipose Tissue in the Progression of Weight Loss After Sleeve Gastrectomy in Morbidly Obese Patients.
Brief Title: Role NLRP3 Inflammasome in Weight Loss Following Sleeve Gastrectomy in Morbidly Obese Patients
Acronym: BARIAMITRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Other Study IDs: 18_RIPH3-14
Record Dates: First submitted 2020-11-24; First posted 2021-03-24 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Obesity Morbid; Obesity-Associated Insulin Resistance
Keywords: Obesity, cardiovascular risk, diabetes
MeSH Terms: conditions — Obesity, Morbid; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Measure of NLRP3 inflammasome preoperative activation level by the expression of NLRP3, IL-1β, IL18 and caspase-1 mRNAs in subcutaneous and visceral adipose tissue. of the epiploon;

SUMMARY:
Epidemiological studies show a very rapid increase in the epidemic of obesity in the Caribbean population. 6 out of 10 adults are overweight and 1 out of 4 is obese. Most are women.

Consequences : harm to health and possible reduction in life expectancy due to the association with many cardiovascular comorbidities.

Adverse effects of obesity on the cardiovascular and endocrine systems are attributed a chronic low-grade inflammatory state in obese patients. Visceral adipose tissue is largely responsible for the inflammatory syndrome. Obesity can also induce the formation of multi-protein platforms called inflammasomes also activated by mitochondrial production.

Morbid obesity treatment with sleeve gastrectomy is an effective long term therapeutic for weight loss but also beneficial in terms of insulin resistance and cardiovascular complications.

Some patients nevertheless remain resistant to the beneficial cardio-metabolic effects of bariatric surgery.

However, the mechanisms that regulate the extent of weight loss and its stabilization after bariatric surgery are still poorly understood.

Our study aims to describe the evolution of postoperative weight loss and the place of preoperative inflammation in its amplitude.

The hypothesis is that the level of inflammation in visceral fat before surgery determines the extent of postoperative weight loss in obese women who have undergone sleeve gastrectomy.

DETAILED DESCRIPTION:
Epidemiological studies show a very rapid increase in the epidemic of obesity in the Caribbean population. The latest prevalence data in Martinique show that 6 out of 10 adults are overweight and 1 out of 4 is obese (Body Mass Index, BMI ≥ 30 kg/m2). Obesity with a BMI ≥ 35 kg/m2 is said to be "morbid" because of its association with numerous cardiovascular comorbidities. A balanced diet and physical activity are effective behavioural modalities for weight loss, which, even at low intensity, can reduce cardiovascular complications and the risk of death. However, many patients do not adhere to these constraints over a long period of time and about 50% of them regain weight after the first year. These observations highlight the value of alternative therapies with lasting effects on weight loss and the cardio-metabolic comorbidities of obesity.

Bariatric surgery with vertical calibrated vertical gastroplasty with gastric resection (or sleeve gastrectomy) and Roux-en-Y gastric bypass are therapeutic options that are not only effective in the long term for weight loss but also beneficial in terms of insulin resistance and cardiovascular complications. Bariatric surgery is currently indicated for the treatment of morbid obesity with a BMI ≥ 40 kg/m2 or a BMI ≥ 35 kg/m2 in the presence of complications. Some patients nevertheless remain resistant to the beneficial cardio-metabolic effects of bariatric surgery. The reasons for this resistance are attributed to factors such as age > 60 years, female sex, BMI > 45 kg/m2, African-American or Hispanic origin, and history of type 2 diabetes. Regardless of these factors, several studies have pointed out that a chronic low-grade inflammatory state reduces the magnitude of weight loss and thus counters the beneficial cardio-metabolic effects of bariatric surgery.

Visceral adipose tissue is largely responsible for the inflammatory syndrome in obese patients, via the activation of nuclear transcription factors (NFkB, in particular) that stimulate the synthesis of numerous mediators and pro-inflammatory cytokines. Obesity can also induce the formation of multi-protein platforms called inflammasomes, including the active assembly of inflammatory caspases (caspase-1, in particular) that cleave the pro-interleukins IL1β and IL18 into mature pro-inflammatory cytokines IL1β and IL18. The role of the inflammasome NLRP3 ("NOD-like receptor family, pyrin domain containing 3") in the inflammatory response has been particularly studied in humans due to its association with multiple chronic inflammatory, infectious and cardio-metabolic pathologies. Among the biomolecules responsible for activation of the NLRP3 inflammasome during obesity are palmitate, sphingolipids and cholesterol crystals. The NLRP3 inflammasome is also activated by mitochondrial production of reactive oxygen species (ROS) and by mitochondrial DNA released from mitochondria damaged by lipo-toxicity phenomena associated with obesity. More generally, the mitochondrial dysfunction of the metabolic syndrome is considered to be the causal intracellular event of the deregulation of the inflammatory response mediated by the inflammasome.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman between the ages of 18 and 45;
* Have been well informed about bariatric surgery and perioperative risks and have benefited from a multidisciplinary evaluation by a multidisciplinary team (RCP) ;
* Have a BMI greater than or equal to 40 kg/m2 or greater than or equal to 35 kg/m2 with at least one co-morbidity that can be improved after surgery (cardiovascular disease, sleep apnea and severe respiratory disorders, type 2 diabetes, osteoarticular diseases)
* Have been informed of the research on the samples taken during care;
* Having stated its decision not to object to the research on the samples taken during the treatment;
* To have accepted medical and surgical follow-up for 24 months;
* Patient under the general social security system.

Exclusion Criteria:

* Being a pregnant or nursing woman;
* Being a type 1 diabetic;
* Have inflammatory bowel disease;
* Have severe and unstable eating disorders ;
* Have severe, uncontrolled cognitive, mental or psychological disorders;
* Have a cancerous pathology;
* Be addicted to alcohol and psychoactive substances (both legal and illegal);
* Have a life-threatening illness in the short or medium term;
* Have contraindications related to surgical operations in general such as general anaesthesia;
* Be under legal protection measures (guardianship, curators, safeguarding of justice), and person deprived of liberty.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Due to the almost exclusive type of recruitment of obese women by the obesity management centre of CHU Martinique (around 90% of patients), only obese women aged between 18 and 45 years old will be included in the study. Only patients who have undergone a sleeve gastrectomy will be included in the study, as this surgical procedure is performed on approximately 9 out of 10 patients in the digestive surgery department of the CHU de Martinique.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-03-13 (Actual); Primary Completion 2024-06-13 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Weight loss (kg) at 12 months of sleeve gastrectomy | 12 months
  Magnitude of weight loss (kg) at 12 months of sleeve gastrectomy as a function of the level of preoperative activation of the NLRP3 inflammasome.

SECONDARY OUTCOMES:
Preoperative activation level of the NLRP3 inflammasome | 1 day
  Preoperative activation level of the NLRP3 inflammasome will be measured by the expression of NLRP3, IL-1β, IL18 and caspase-1 mRNAs in subcutaneous and visceral adipose tissue of the epiploon; expressed as mRNA copy number measured in quantitative RT-PCR (RT-qPCR)
Mitochondrial activity | 1 day
  Preoperative levels of oxygen consumption by the mitochondrial respiratory chain (pmol O2*s-1*mg-1 of dry tissue)
Pre and post operative inflammatory state | 24 months
  Pre- and post-operative plasma levels of CRP and proinflammatory cytokines IL-1β and IL18 (pg/mL). Postoperative measurements will be done up to 6 months after bariatric surgery. In addition, since fat tissue sampling is not justified postoperatively, activation of the NLRP3 inflammasome will be assessed indirectly by plasma concentrations of the cytokines IL-1β and IL18
Pre and post-operative BMI | 24 months
  Weight and height will be combined to report BMI in kg/m^2) at pre- and post-operative
Pre and post-operative abdominal perimeter | 24 months
  Abdominal perimeter in centimeter at pre- and post-operative (24-month follow-up).
Pre and post-operative hip circumference | 24 months
  Hip circumference in centimeter at pre- and post-operative (24-month follow-up).

CONTACTS AND LOCATIONS:
Overall Officials: Rémi NEVIERE, MD, PhD, Study Chair — CHU de Martinique; Emmanuel RIVKINE, Principal Investigator — CHU de Martinique
Locations (1):
- CHU de Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neeland IJ, Poirier P, Despres JP. Cardiovascular and Metabolic Heterogeneity of Obesity: Clinical Challenges and Implications for Management. Circulation. 2018 Mar 27;137(13):1391-1406. doi: 10.1161/CIRCULATIONAHA.117.029617. PMID 29581366
- [Result] Vecchie A, Dallegri F, Carbone F, Bonaventura A, Liberale L, Portincasa P, Fruhbeck G, Montecucco F. Obesity phenotypes and their paradoxical association with cardiovascular diseases. Eur J Intern Med. 2018 Feb;48:6-17. doi: 10.1016/j.ejim.2017.10.020. PMID 29100895
- [Result] le Roux CW, Heneghan HM. Bariatric Surgery for Obesity. Med Clin North Am. 2018 Jan;102(1):165-182. doi: 10.1016/j.mcna.2017.08.011. PMID 29156184
- [Result] Pareek M, Schauer PR, Kaplan LM, Leiter LA, Rubino F, Bhatt DL. Metabolic Surgery: Weight Loss, Diabetes, and Beyond. J Am Coll Cardiol. 2018 Feb 13;71(6):670-687. doi: 10.1016/j.jacc.2017.12.014. PMID 29420964
- [Result] Lupoli R, Lembo E, Saldalamacchia G, Avola CK, Angrisani L, Capaldo B. Bariatric surgery and long-term nutritional issues. World J Diabetes. 2017 Nov 15;8(11):464-474. doi: 10.4239/wjd.v8.i11.464. PMID 29204255
- See also: WHO : obesity and overweight — http://www.who.int/fr/news-room/fact-sheets/detail/obesity-and-overweight
- See also: Overweight and abdominal obesity (KANNARI study in Martinique) — https://www.martinique.ars.sante.fr/system/files/2018-03/4%20pages%20Kannari%20OSM_surcharge%20pondérale%20%282%29.pdf